CLINICAL TRIAL: NCT01161160
Title: An Observer-blind Safety and Immunogenicity Study of GSK Biologicals' A/California/7/2009 (H1N1)V-like Vaccines GSK2340274A and GSK2340272A in Children 3 to Less Than 10 Years Old
Brief Title: Safety and Immune Response of Candidate H1N1 Influenza Vaccines GSK2340274A and GSK234072A in Children 3 to Less Than 10 Years Old
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 114495
Record Dates: First submitted 2010-07-01; First posted 2010-07-13 (Estimated); Results first posted 2017-08-04 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2017-04

CONDITIONS: Influenza
Keywords: H1N1; Influenza; Pandemic; GSK Bio's influenza vaccines GSK2340274A and GSK234072A
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- AREPANRIX 1/2 GROUP (Experimental): Healthy male or female children aged 3 to less than (<) 10 years at the time of study vaccination, who received 1 half (1/2) pediatric dose of Arepanrix™ vaccine at Day 0, administered intramuscularly in the deltoid of the non-dominant arm.
  Interventions: Biological: GSK Biologicals' GSK2340274A (two different formulations)
- PANDEMRIX 1/2 GROUP (Experimental): Healthy male or female children aged 3 to less than (<) 10 years at the time of study vaccination, who received 1 half (1/2) pediatric dose of Pandemrix™ vaccine at Day 0, administered intramuscularly in the deltoid of the non-dominant arm.
  Interventions: Biological: GSK Biologicals' - GSK2340272A
- AREPANRIX GROUP (Experimental): Healthy male or female children aged 3 to less than (<) 10 years at the time of study vaccination, who received 1 pediatric dose of Arepanrix™ vaccine at Day 0, administered intramuscularly in the deltoid of the non-dominant arm.
  Interventions: Biological: GSK Biologicals' GSK2340274A (two different formulations)

INTERVENTIONS:
Biological: GSK Biologicals' GSK2340274A (two different formulations) — Intramuscular injection
  Arms: AREPANRIX 1/2 GROUP; AREPANRIX GROUP
Biological: GSK Biologicals' - GSK2340272A — Intramuscular injection
  Arms: PANDEMRIX 1/2 GROUP

SUMMARY:
This study is designed to characterize the safety and immunogenicity of pandemic influenza (H1N1) candidate vaccines GSK2340274A and GSK234072A in children 3 to less than 10 years old.

ELIGIBILITY:
Inclusion Criteria:

* Male or pre-menarchal female children 3 to < 10 years of age at the time of the study vaccination. "Less than 10 years of age" implies inclusion of children who have not reached their 10th birthday as of Day 0, the day of the study vaccine dose under this protocol.
* Written informed consent obtained from the subject's parent/legally acceptable representative (LAR); written informed assent obtained from the subject if appropriate.
* Good general health as established by medical history and clinical examination before entering into the study.
* Subjects and/or parent(s)/LAR who the investigator believes can and will comply with the requirements of the protocol as documented by signature on the informed consent document (and, if appropriate, the informed assent document).

Exclusion Criteria:

* Medical history of physician-confirmed infection with an A/California/7/2009 (H1N1)v-like virus.
* Previous vaccination at any time with an A/California/7/2009 (H1N1)v-like virus vaccine.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, even if stable, are deemed by the investigator to render the potential subject or parent(s)/ LAR(s) unable/unlikely to provide accurate safety reports.
* Presence of a temperature ≥ 38.0ºC by any route or method, or acute symptoms greater than "mild" severity on the scheduled date of vaccination.
* Diagnosed with cancer, or treatment for cancer, within 3 years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Receipt of systemic glucocorticoids within 1 month prior to study enrollment (day of study vaccination), or any other cytotoxic or immunosuppressive drug within 6 months of study enrollment. Topical, intra-articular or inhaled glucocorticoids are allowed.
* Receipt of any immunoglobulins and/or any blood products within 6 months of study enrollment or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin are eligible if no such doses are given in the 24 hours before a study vaccination. Persons receiving prophylactic antiplatelet medications, e.g., low-dose acetylsalicylic acid, and without a clinically-apparent bleeding tendency, are eligible.
* Administration of any licensed live-attenuated vaccine within 30 days before study vaccination or any licensed inactivated vaccine within 15 days before study vaccination.
* Planned administration of any A/California H1N1v-like vaccine other than the study vaccine between Day 0 and the Day 21 phlebotomy.
* Planned administration of any other vaccine not foreseen by the study protocol between Day 0 and Day 21. Routine childhood vaccinations are exempted if they cannot be delayed, but they must not be administered on the same day as the H1N1 vaccine candidate.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding study vaccination, or planned use during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Child in care (A child who has been placed under the control or protection of an agency, organization, institution or entity by the courts).

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 209 (Actual)
Dates: Start 2010-07-01; Primary Completion 2010-08-23 (Actual); Study Completion 2011-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Sampaloc, Manila, Philippines
- GSK Investigational Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Launay O, Duval X, Fitoussi S, Jilg W, Kerdpanich A, Montellano M, Schwarz TF, Watanveerade V, Wenzel JJ, Zalcman G, Bambure V, Li P, Caplanusi A, Madan A, Gillard P, Vaughn DW. Extended antigen sparing potential of AS03-adjuvanted pandemic H1N1 vaccines in children, and immunological equivalence of two formulations of AS03-adjuvanted H1N1 vaccines: results from two randomised trials. BMC Infect Dis. 2013 Sep 16;13:435. doi: 10.1186/1471-2334-13-435. PMID 24041010
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 114495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Period: Overall Study
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Started | 76 | 75 | 58
Completed | 76 | 75 | 58
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group | Total
Number analyzed (Participants) | 76 | 75 | 58 | 209
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6 (2.03) | 6 (2.02) | 6 (2) | 6 (2.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 38 | 27 | 95
  Male | 46 | 37 | 31 | 114
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-Central/South Asian heritage | 0 | 1 | 0 | 1
  Asian-East Asian heritage | 0 | 0 | 1 | 1
  Asian-South East Asian heritage | 76 | 74 | 57 | 207

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects for Haemagglutination Inhibition (HI) Antibodies Against Flu A/CAL/7/09 H1N1 Strain
Description: Seroconversion rate (SCR) was defined as the proportion of subjects who had either a pre-vaccination reciprocal HI titer below (<) 10 and a post-vaccination reciprocal titre greater than or equal to (≥) 40, or a pre-vaccination reciprocal HI titer ≥ 10 and at least a 4-fold increase in post vaccination reciprocal titer against the vaccine virus. The Flu strain assessed was A/California/7/2009 (H1N1)v-like virus (Flu A/CAL/7/09), following the Committee for Medicinal Products for Human Use (CHMP) and the Center for Biologics Evaluation and Research (CBER) guidance. The CBER criterion was fulfilled if the lower 95% confidence interval (CI) for SCR was (>) 40%. The CHMP criterion was fulfilled if the point estimate for SCR was > 40%.
Time Frame: At Day 21
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity at Day 21, which included all evaluable subjects for whom assay results for antibodies against A/California-like HA antigen for the blood sample taken 21 days after vaccination were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 76 | 75 | 58
Participants | 75 | 74 | 57

2. Primary Outcome: Number of Seroprotected Subjects for HI Antibodies Against Flu A/CAL/7/09 H1N1 Strain
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40, that usually is accepted as indicating protection. The Flu strain assessed was Flu A/CAL/7/09, following the CHMP and the CBER guidance. The CBER criterion was fulfilled if the lower limit of the 95% CI for seroprotection (SPR) was > 70%. The CHMP criterion was fulfilled if the post-vaccination point estimate for SPR was > 70%.
Time Frame: At Day 0
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 21, which included all evaluable subjects for whom assay results for antibodies against A/California-like HA antigen for the blood sample taken 21 days after vaccination were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 76 | 75 | 58
Participants | 28 | 24 | 18

3. Primary Outcome: Number of Seroprotected Subjects for HI Antibodies Against Flu A/CAL/7/09 H1N1 Strain
Description: as for outcome 2
Time Frame: At Day 21
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 21, which included all evaluable subjeects for whom assay results for antibodies against A/California-like HA antigen for the blood sample taken 21 days after vaccination were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 76 | 75 | 58
Participants | 75 | 74 | 57

4. Primary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/CAL/7/09 H1N1 Strain
Description: GMFR, also called seroconversion factor (SCF), was defined as the fold increase in serum HI geometric mean titers (GMTs) post-vaccination compared to pre-vaccination. The Flu strain assessed was Flu A/CAL/7/09, following the CHMP and the CBER guidance. The CHMP criterion was fulfilled if the point estimate for GMFR was > 2.5.
Time Frame: At Day 21
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 76 | 75 | 58
Fold increase | 25.7 [20.7 to 32] | 27.1 [22.4 to 32.8] | 32.2 [24.7 to 42.0]

5. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies Against Flu A/CAL/7/09 H1N1 Strain
Description: Seroconversion rate (SCR) was defined as the proportion of subjects who had either a pre-vaccination reciprocal HI titer < 10 and a post-vaccination reciprocal titer ≥ 40, or a pre-vaccination reciprocal HI titer ≥ 10 and at least a 4-fold increase in post vaccination reciprocal titer against the vaccine virus. The Flu strain assessed was Flu A/CAL/7/09, following the CHMP and the CBER guidance. The CBER criterion was fulfilled if the lower limit of the 95% CI for SCR was > 40%. The CHMP criterion was fulfilled if the post-vaccination point estimate for SCR was > 40%.
Time Frame: At Day 182
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 182, which included all evaluable subjects for whom assay results for antibodies against A/California-like HA antigen for the blood sample taken 182 days after vaccination were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 73 | 74 | 58
Participants | 46 | 53 | 40

6. Secondary Outcome: Number of Seroprotected Subjects for HI Antibodies Against Flu A/CAL/7/09 H1N1 Strain
Description: as for outcome 2
Time Frame: At Day 0 and Day 182
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 73 | 74 | 58
Participants
  Flu A/CAL/7/09, Day 0 | 27 | 24 | 18
  Flu A/CAL/7/09, Day 182 | 55 | 63 | 46

7. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/CAL/7/09 H1N1 Strain
Description: GMFR, also called seroconversion factor (SCF), was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination. The Flu strain assessed was Flu A/CAL/7/09, following the CHMP and the CBER guidance. The CHMP criterion was fulfilled if the post-vaccination point estimate for SCF was > 2.5.
Time Frame: At Day 182
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 73 | 74 | 58
Fold increase | 6.6 [5.4 to 8.2] | 8 [6.4 to 10.1] | 8.9 [6.8 to 11.7]

8. Secondary Outcome: Number of Subjects With HI Antibody Titers Against Flu A/CAL/7/09 H1N1 Above the Cut-off Value
Description: The cut-off value for the humoral immune response in terms of vaccine H1N1 HI antibodies were egual to or above (≥) 1:10. The Flu strain assessed was Flu A/CAL/7/09, following the CHMP and the CBER guidance.
Time Frame: At Day 21
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 76 | 75 | 58
Participants | 76 | 75 | 58

9. Secondary Outcome: HI Antibody Titers Against Flu A/CAL/7/09 H1N1 Strain
Description: Titers are presented as geometric mean titers (GMTs), for the seropositivity cut-off value of ≥ 1:10. The Flu strain assessed was Flu A/CAL/7/09, following the CHMP and the CBER guidance.
Time Frame: At Day 21
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 76 | 75 | 58
Titers | 448.6 [323.9 to 621.3] | 434.1 [321 to 587] | 418.8 [297.6 to 589.1]
Statistical Analysis 1: Comparison: Arepanrix 1/2 Group vs Pandemrix 1/2 Group; To demonstrate the immunological equivalence of HA antigen adjuvanted with AS03B manufactured in Quebec (Arepanrix™) and HA antigen adjuvanted with AS03B manufactured in Dresden (Pandemrix™), 21 days after vaccination; Test type: Non-Inferiority — Equivalence criteria were fulfilled if the 2-sided 95% confidence limits on the geometric mean titer (GMT) ratio was within the interval 0.5 to 2.0; Adjusted GMT ratio = 0.96, 95% CI 2-sided [0.73 to 1.26]

10. Secondary Outcome: Number of Subjects With HI Antibody Titers Against Flu A/CAL/7/09 H1N1 Above the Cut-off Value
Description: The cut-off value for the humoral immune response in terms of vaccine H1N1 HI antibodies were equal to or above (≥) 1:10. The Flu strain assessed was Flu A/CAL/7/09, following the CHMP and the CBER guidance.
Time Frame: At Day 182
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 73 | 74 | 58
Participants | 72 | 72 | 58

11. Secondary Outcome: HI Antibody Titers Against Flu A/CAL/7/09 H1N1 Strain
Description: Titers were presented as geometric mean titers (GMTs), for the seropositivity cut-off value of ≥ 1:10. The Flu strain assessed was Flu A/CAL/7/09, following the CHMP and the CBER guidance.
Time Frame: At Day 182
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 73 | 74 | 58
Titers | 117.4 [84.5 to 163.1] | 128.3 [95.8 to 171.9] | 115.7 [80.7 to 166]

12. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of any local symptom regardless of intensity grade. Grade 3 pain for children less than 6 years= cried when limb was moved/spontaneously painful. Grade 3 pain for children aged 6 to < 10 years= pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects who received the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 76 | 75 | 58
Participants
  Any Pain | 41 | 41 | 23
  Grade 3 Pain | 3 | 0 | 0
  Any Redness | 0 | 1 | 0
  Grade 3 Redness | 0 | 0 | 0
  Any Swelling | 1 | 5 | 1
  Grade 3 Swelling | 0 | 0 | 0

13. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and fever [defined as axillary temperature equal to or above 38.0 degrees Celsius (°C)]. Any = occurrence of any general symptom regardless of intensity grade or relation to vaccination. Grade 3 drowsiness= drowsiness that prevented normal activity. Grade 3 irritability= crying that could not be comforted/prevented normal activity. Grade 3 loss of appetite= not eating at all. Grade 3 fever = fever > 39.0 °C or > 40.0 °C. Related= general symptom assessed by the investigator as causally related to the vaccination. This outcome measure refers to subjects aged 3 to 5 years.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects aged 3 to 5 years who received the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 33 | 31 | 24
Participants
  Any Drowsiness | 5 | 3 | 1
  Grade 3 Drowsiness | 0 | 0 | 0
  Related Drowsiness | 1 | 2 | 0
  Any Irritability | 2 | 7 | 1
  Grade 3 Irritability | 0 | 0 | 0
  Related Irritability | 0 | 2 | 0
  Any Loss of appetite | 6 | 4 | 1
  Grade 3 Loss of appetite | 1 | 1 | 0
  Related Loss of appetite | 1 | 2 | 0
  Any Fever | 2 | 5 | 5
  Grade 3 Fever | 1 | 2 | 1
  Related Fever | 1 | 5 | 2

14. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms, headache, joint pain at other location, muscle aches, shivering, sweating and fever [defined as axillary temperature equal to or above 38.0 degrees Celsius (°C)]. Any = occurrence of any general symptom regardless of intensity grade or relation to vaccination. Grade 3 symptom= symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C, but ≤ 40.0 °C. Related= general symptom assessed by the investigator as causally related to the vaccination. This outcome measure refers to subjects aged 6 to 10 years.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects aged 6 to 10 years who received the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 41 | 44 | 33
Participants
  Any Fatigue | 4 | 3 | 2
  Grade 3 Fatigue | 1 | 0 | 0
  Related Fatigue | 1 | 0 | 0
  Any Gastrointestinal | 2 | 1 | 0
  Grade 3 Gastrointestinal | 1 | 0 | 0
  Related Gastrointestinal | 0 | 0 | 0
  Any Headache | 7 | 9 | 4
  Grade 3 Headache | 1 | 0 | 0
  Related Headache | 0 | 2 | 0
  Any Joint pain at other location | 5 | 1 | 4
  Grade 3 Joint pain at other location | 1 | 0 | 0
  Related Joint pain at other location | 1 | 0 | 0
  Any Muscle aches | 6 | 7 | 5
  Grade 3 Muscle aches | 0 | 0 | 0
  Related Muscle aches | 1 | 1 | 0
  Any Shivering | 4 | 2 | 0
  Grade 3 Shivering | 1 | 0 | 0
  Related Shivering | 0 | 0 | 0
  Any Sweating | 2 | 1 | 0
  Grade 3 Sweating | 1 | 0 | 0
  Related Sweating | 0 | 0 | 0
  Any Fever | 4 | 0 | 0
  Grade 3 Fever | 1 | 0 | 0
  Related Fever | 1 | 0 | 0

15. Secondary Outcome: Number of Subjects With Medically-attended Adverse Events (MAEs)
Description: MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any MAE(s) = Occurrence of any MAE(s) regardless of intensity grade or relation to vaccination. Analysis of intensity and relationship to vaccination of MAEs was not performed.
Time Frame: Up to day 21
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects who received the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 76 | 75 | 58
Participants | 14 | 9 | 1

16. Secondary Outcome: Number of Subjects With MAEs
Description: as for outcome 15
Time Frame: During the entire study period (Day 0 to Day 182)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects who received the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 76 | 75 | 58
Participants | 29 | 29 | 18

17. Secondary Outcome: Number of Subjects With Potential Immune-mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: Up to Day 21
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects who received the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 76 | 75 | 58
Participants | 0 | 0 | 0

18. Secondary Outcome: Number of Subjects With pIMDs
Description: as for outcome 17
Time Frame: During the entire study period (Day 0 to Day 182)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects who received the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 76 | 75 | 58
Participants | 0 | 0 | 0

19. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within the 21-day (Days 0-20) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects who received the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 76 | 75 | 58
Participants | 22 | 21 | 5

20. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: as for outcome 19
Time Frame: Within the 42-day (Days 0-41) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects who received the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 76 | 75 | 58
Participants | 28 | 28 | 23

21. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Up to 21 days after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects who received the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 76 | 75 | 58
Participants | 0 | 0 | 0

22. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 19
Time Frame: During the entire study period (Day 0 to Day 182)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects who received the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
Number analyzed (Participants) | 76 | 75 | 58
Participants | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicted AEs: during the 42-day (Days 0-41) post-vaccination period; SAEs: during the entire study period (from Day 0 up to Day 182).
Description: The solicited local and general symptoms were only collected for those subjects who filled in their symptom sheets.
Arm/Group | Arepanrix 1/2 Group | Pandemrix 1/2 Group | Arepanrix Group
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/75 | 0/58
Serious Adverse Events (participants affected / at risk) | 1/76 | 0/75 | 1/58
Other Adverse Events (participants affected / at risk) | 52/76 | 52/75 | 35/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arepanrix 1/2 Group (N=76) | Pandemrix 1/2 Group (N=75) | Arepanrix Group (N=58)
Dengue fever (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Arepanrix 1/2 Group (N=76) | Pandemrix 1/2 Group (N=75) | Arepanrix Group (N=58)
Cough (Days 0-41 post-vacc.) (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3
Conjunctivitis (Days 0-41 post-vacc.) (Eye disorders) | 3 | 1 | 3
Pyrexia (Days 0-20 post-vacc.) (General disorders) | 2 | 6 | 1
Pyrexia (Days 0-41 post-vacc.) (General disorders) | 4 | 9 | 6
Pain (General disorders) | 41 | 41 | 23
Swelling (General disorders) | 1 | 5 | 1
Drowsiness (3-5Y) (General disorders) | 5/33 | 3/31 | 1/24
Irritability (3-5Y) (General disorders) | 2/33 | 7/31 | 1/24
Loss of appetite (3-5Y) (General disorders) | 6/33 | 4/31 | 1/24
Temperature/Axillary (3-5Y) (General disorders) | 2/33 | 5/31 | 5/24
Fatigue (6-10Y) (General disorders) | 4/41 | 3/44 | 2/33
Headache (6-10Y) (General disorders) | 7/41 | 9/44 | 4/33
Joint pain (6-10Y) (General disorders) | 5/41 | 1/44 | 4/33
Muscle aches (6-10Y) (General disorders) | 6/41 | 7/44 | 5/33
Shivering (6-10Y) (General disorders) | 4/41 | 2/44 | 0/33
Temperature/Axillary (6-10Y) (General disorders) | 4/41 | 0/44 | 0/33
Upper respiratory tract infection (Days 0-20 post-vacc.) (Infections and infestations) | 5 | 5 | 1
Nasopharyngitis (Days 0-20 post-vacc.) (Infections and infestations) | 5 | 1 | 2
Rhinitis (Days 0-20 post-vacc.) (Infections and infestations) | 4 | 2 | 0
Nasopharyngitis (Days 0-41) (Infections and infestations) | 7 | 5 | 5
Upper respiratory tract infection (Days 0-41 post-vacc.) (Infections and infestations) | 6 | 6 | 3
Rhinitis (Days 0-41 post-vacc.) (Infections and infestations) | 5 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.